CLINICAL TRIAL: NCT00698412
Title: The Impact of Daily Cane Use on Pain, Function, Quality of Life and Energy Consumption During the Gait in Patients With Knee Osteoarthritis
Brief Title: Effectiveness of Cane in Osteoarthritis (OA) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Anamaria Jones, UNIFESP - Universidade Federal de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIFESP-102/2004
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-05

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Daily cane use; Pain; Function; Quality of life; Energy consumption during the gait
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Canes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cane group
  Interventions: Device: Cane
- 2 (No Intervention): Control Group

INTERVENTIONS:
Device: Cane — This group use the cane every day since the baseline
  Arms: 1

SUMMARY:
Sixty four participants were enrolled in a randomized, controlled clinical trial to evaluate the effectiveness of daily cane use on pain, function, quality of life and energy consumption during the gait in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Treatment, Randomized, Single Blind, Parallel Assignment, Efficacy Study

ELIGIBILITY:
Inclusion Criteria:

* Primary Knee osteoarthritis (ACR criteria)
* VAS for knee pain between 3 and 7
* No changes the NSAID intake or physical activity in the previous 3 months

Exclusion Criteria:

* Symptomatic heart or pulmonary disease
* Severe systemic disease
* Other symptomatic disease in the lower limb or in the upper limb that will carry the cane
* Joint injection in the previous 3 months
* PT in the previous 3 months
* Previously cane use
* Start regular physical activity in the last month

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pain - visual analogue scale | T0, T30 and T60

SECONDARY OUTCOMES:
Function - Lequesne index | T0, T30 and T60
Function - WOMAC questionnaire | T0,T30 and T60
Quality of life - SF-36 | T0, T30 and T60
Energy consumption (VO2)- gas analysis with and without cane during the 6MWT | T0, T30 and T60

CONTACTS AND LOCATIONS:
Overall Officials: Anamaria Jones, PT, Principal Investigator — Federal University of São Paulo; Jamil Natour, MD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Jones A, Silva PG, Silva AC, Colucci M, Tuffanin A, Jardim JR, Natour J. Impact of cane use on pain, function, general health and energy expenditure during gait in patients with knee osteoarthritis: a randomised controlled trial. Ann Rheum Dis. 2012 Feb;71(2):172-9. doi: 10.1136/ard.2010.140178. Epub 2011 Nov 29. PMID 22128081